CLINICAL TRIAL: NCT00409383
Title: A Pilot Study of Abraxane® (Albumin-bound Paclitaxel) and Temodar® (Temozolomide) Plus Genasense® (Oblimersen Sodium) in Subjects With Advanced Melanoma ("The ATG Study").
Brief Title: Abraxane and Temodar Plus Genasense in Advanced Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GM108
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2010-07

CONDITIONS: Melanoma
Keywords: Advanced Melanoma; Normal baseline LDH; Chemotherapy naive
MeSH Terms: conditions — Melanoma | interventions — oblimersen; Albumin-Bound Paclitaxel; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Genasense® (oblimersen) — Cohorts 1 and 2: Genasense 7 mg/kg/day by continuous intravenous infusion beginning on Day 1 and continuing for 7 days (Week 1) and beginning again on Day 22 and continuing for 7 days (Week 4); Cohort 3: Genasense 900 mg as a 1-hour intravenous infusion on Day 1, 4, 8, and 11 (Weeks 1 and 2) and Day 22, 25, 29, and 32 (Weeks 4 and 5).
  Other Names: G3139
Drug: Abraxane® (paclitaxel protein-bound particles for injectable suspension) — Cohorts 1 and 2: Abraxane 175 mg/m2 or 260 mg/m2 as a 30-minute intravenous infusion on Day 8 and Day 29 following end of Genasense continuous infusion; Cohort 3: Abraxane 175 mg/m2 as a 30-minute intravenous infusion on Day 4 and Day 25 following end of Genasense 1-hour infusion
  Other Names: albumin-bound paclitaxel
Drug: Temodar® (temozolomide) — Cohorts 1-3: Temodar 75 mg/m2/day orally on Days 1 through 42 (Week 1 through Week 6)

SUMMARY:
This study is designed to evaluate the safety, efficacy, pharmacokinetics, and pharmacodynamics of combination treatment with Temodar®, Genasense®, and Abraxane® in chemotherapy-naïve subjects with advanced melanoma and normal lactate dehydrogenase (LDH).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with progressive, unresectable, or advanced melanoma who are considered to be candidates for systemic treatment with chemotherapy
* Subjects will have measurable disease, an Eastern Cooperative Oncology Group Performance Status less than or equal to 2, and serum LDH less than or equal to 1.1 times the upper limit of normal, but will not have previously received cytotoxic chemotherapy
* Prior immunotherapy, radiotherapy, or cytokine, biologic, or vaccine therapy is permitted in the adjuvant and/or metastatic setting

Exclusion Criteria:

* Prior treatment with cytotoxic chemotherapy, including regional perfusion, or with Genasense®(oblimersen sodium)Injection
* Nonmeasurable disease only
* History or presence of brain metastasis or leptomeningeal disease
* Significant medical disease other than cancer
* Known human immunodeficiency virus infection
* Pregnant or lactating
* Known hypersensitivity to temozolomide, phosphorothioate-containing oligonucleotides, or products containing human albumin
* Use of any experimental therapy within 3 weeks prior to baseline evaluations, Other anticancer treatment (such as chemotherapy, radiation, or biologic or investigational therapies) while receiving therapy in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2006-11; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Safety based on adverse event reports and clinical laboratory findings | During protocol therapy prior to the start of and during each cycle and up to 30 days after last dose of protocol therapy

SECONDARY OUTCOMES:
Response rate (including rate of complete response) | At the end of each cycle during protocol therapy, with follow-up every 2 months for up to 2 years from date of registration
Duration of response (including the rate of durable response) | At the end of each cycle during protocol therapy, with follow-up every 2 months for up to 2 years from date of registration
Time to disease progression | At the end of each cycle during protocol therapy, with follow-up every 2 months for up to 2 years from date of registration
Incidence of brain metastasis | At the end of each cycle during protocol therapy, with follow-up every 2 months for up to 2 years from date of registration
Survival | 12,15, and 18 months from date of registration, with follow-up every 2 months for up to 2 years from date of registration
Correlations of drug concentrations, intracellular Bcl-2 content, and response | Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Anna C Pavlick, MD, Principal Investigator — NYU MEDICAL CENTER
Locations (1):
- New York University Cancer Center, New York, New York, United States